CLINICAL TRIAL: NCT03187652
Title: A Prospective Study on the Long-Term Vascular Burden in Thrombotic Thrombocytopenic Purpura Patients
Acronym: TTP
Status: Recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 108273
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT Perfusion Study — Brain and cardiac CT perfusion scan
Diagnostic Test: Echocardiogram — Speckle tracking Echocardiography
Diagnostic Test: neuro-cognitive assessment — Cambridge Brain Sciences neuro-cognitive assessment
Diagnostic Test: MRI — MRI to assess white matter changes

SUMMARY:
A prospective cohort study of thrombotic thrombocytopenic purpura and atypical hemolytic uremic syndrome patients who have presented with their acute episode and are in remission within the last 30 days. They will be followed for 12 months from the time of their initial scan, followed by a long-term follow up study.

DETAILED DESCRIPTION:
The investigators will conduct a prospective cohort study at the London Health Sciences Centre, Ontario, Canada. The investigators will identify 15-30 idiopathic thrombotic thrombocytopenic purpura and atypical hemolytic uremic syndrome patients who are in remission within the last 30 days. They will be followed for 12 months from the time of their remission. Study procedures include routine laboratory monitoring, biomarker assessments, cardiovascular and neurocognitive functional assessments, and non-invasive imaging studies. The long-term follow-up thrombotic thrombocytopenic purpura and atypical hemolytic uremic syndrome study will help to assess the mechanisms of vascular injuries, evaluate cardiovascular and cerebrovascular monitoring tools, and generate novel ideas to prevent further vascular injuries.

ELIGIBILITY:
Inclusion Criteria:

* Adults (=18 years) with a recent diagnosis of their first episode of idiopathic TTP, who have been treated with plasma exchange with or without other therapies, and who are in remission. Remission is defined as the normalization of platelet counts and lactate dehydrogenase levels with no clinical signs or symptoms of microvascular injury for more than 30 days. The patients will be included in the study within 30 days of remission of their symptoms. The patients will all meet the following diagnostic criteria for idiopathic TTP: (1) thrombocytopenia with platelet count <150 x 109 /L, (2) microangiopathic hemolytic anaemia (presence of red blood cell fragmentation by peripheral blood smear), (3) elevation of lactate dehydrogenase (LDH)> 1.25 X of the upper limit of normal, and (4) ADAMTS13 Activity < 10%

Exclusion Criteria:

* Patients will be excluded if they have diagnoses of typical HUS (diarrhea-associated HUS), atypical HUS, and disseminated intravascular coagulation, have abnormal international normalized ratio at the time of presentation, have diagnoses of malignant hypertension at the time of presentation, are on the following drugs within 90 days prior to their presentation: ticlopidine, clopidogrel, mitomycin C, gemcitabine, cyclosporine, and quinine, have a history of hematopoietic stem cell transplantations prior to their presentation, have a history and/or diagnosis of vasculitis, systemic lupus erythematosus, scleroderma, rheumatoid arthritis, antiphospholipid antibody syndrome, or HIV/AIDS, have a history of solid organ malignancy within 5 years prior to presentation, i.e. lung, breast, gastric, colon, pancreatic, prostate, or liver, are pregnant at the time of presentation, have severe bronchospasm, unstable angina, and severe ischemic heart disease, have advanced kidney failure (estimated Glomerular Filtration Rate < 30 mL/min/1.73m2), and have history of allergic reaction to contrast dye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic TTP
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
vascular events affecting the brain and heart | 0-12 months
  The investigators will report the proportion of patients who have functional and/or structural vascular events affecting the brain and heart, after the first acute idiopathic TTP events

CONTACTS AND LOCATIONS:
Overall Officials: Huang, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hannan F, Hamilton J, Patriquin CJ, Pavenski K, Jurkiewicz MT, Tristao L, Owen AM, Kosalka PK, Deoni SCL, Theberge J, Mandzia J, Huang SHS, Thiessen JD. Cognitive decline in thrombotic thrombocytopenic purpura survivors: The role of white matter health as assessed by MRI. Br J Haematol. 2024 Mar;204(3):1005-1016. doi: 10.1111/bjh.19246. Epub 2023 Dec 11. PMID 38083818